CLINICAL TRIAL: NCT06407661
Title: How Does the Disaster Nursing Course Affect Nursing Students' Disaster Literacy and Preparedness Perceptions?
Brief Title: Disaster Nursing Course Affect Nursing Students' Disaster Literacy and Preparedness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Özüm Erkin, Associate Professor, Izmir Democracy University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IDU-SBF-ÖE-02
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Literacy
Keywords: literacy; nursing student
MeSH Terms: conditions — Literacy | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The study was a one-group quasi-experimental study design in a pretest-posttest design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental): In this study, the "Disaster Nursing" course, which was integrated into the nursing curriculum, was an elective course, and it was carried out as a theoretical course for two hours a week. The purpose of its development was to educate students on disaster management and disaster nursing [54]. The course content included identification of risks and resources for disasters at the primary protection level, nurse's caregiver (triage and holistic care) and case manager role at the secondary protection level, reassessment of individuals' care needs at the tertiary level, and review of education and the current disaster plan at the protection level. The disaster nursing course was intended to develop students' perception of disaster awareness, preparedness, and response self-efficacy by providing them with primary, secondary, and tertiary level protection roles
  Interventions: Other: "Disaster Nursing" course/education

INTERVENTIONS:
Other: "Disaster Nursing" course/education — In this study, the "Disaster Nursing" course, which was integrated into the nursing curriculum, was an elective course, and it was carried out as a theoretical course for two hours a week. The topics in the content of this course regarding prevention, preparedness, response and recovery stages were designed in line with Jennings Disaster Nursing Management Model. The purpose of its development was to educate students on disaster management and disaster nursing. The course content included identification of risks and resources for disasters at the primary protection level, nurse's caregiver (triage and holistic care) and case manager role at the secondary protection level, reassessment of individuals' care needs at the tertiary level, and review of education and the current disaster plan at the protection level.

SUMMARY:
This study aimed to examine the effect of disaster nursing course on nursing students' disaster literacy and preparedness perceptions. The study, which was a one-group quasi-experimental study design in a pretest-posttest design. Pre-test was done on September 27, 2021, and the post-test was applied on January 7, 2022. The location of the study is a public university in Izmir which is located in western part of Türkiye. The population of the study consisted of nursing students (n: 66) studying in the nursing department of the university and enrolled in the elective course "Disaster Nursing". No sample selection was made, and the study was conducted with 62 volunteer students. Individual introduction form, Disaster Literacy Scale, and Perception of Disaster Preparedness in Nurses Scale were used as tools for data collection. At the beginning of the study, data collection tools were collected online form. "Disaster nursing" course was conducted for 14 weeks as an intervention. The data were stored in the SPSS 25 program.

DETAILED DESCRIPTION:
This study aimed to examine the effect of disaster nursing course on nursing students' disaster literacy and preparedness perceptions. The study was a one-group quasi-experimental study design in a pretest-posttest design. Pre-test was done on September 27, 2021, and the post-test was applied on January 7, 2022. The location of the study is a public university in Izmir which is located in the western part of Türkiye. The population of the study consisted of nursing students (n: 66) studying in the nursing department of the university and enrolled in the elective course "Disaster Nursing". No sample selection was made, and the study was conducted with 62 volunteer students. Individual introduction form (13 questions), Disaster Literacy Scale (61 items), and Perception of Disaster Preparedness in Nurses Scale (20 items) were used as tools for data collection. At the beginning of the study, data collection tools were collected online form. "Disaster nursing" course was conducted for 14 weeks as an intervention. The descriptive statistical methods (number, percentage, mean, standard deviation), paired sample t-test, and Pearson correlation was used data analysis.

ELIGIBILITY:
Inclusion Criteria:

* enrollment in the disaster nursing course
* regular attendance at meetings
* voluntary participation in the study

Exclusion Criteria:

* participants with any form of cognitive
* a mental, or physical disability that interfered with communication,
* as well as individuals with an employment history, a diploma, or a certificate in the subject of disaster

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Disaster Literacy Scale (DLS) | 14 weeks
  The conceptual framework of the 61-item scale consists of 16 domains.There are no reverse coded items in the scale. For ease of score calculation, the total score was standardized in the range of 0-50: Formula = Index = (arithmetic mean - 1) x [50/4]. With the calculated formula, cut-off points for harm reduction, preparedness, response and recovery dimensions were determined by SS values based on z-score. On the scale, 0 represents the lowest DLS and 50 represents the highest DLS. "The scale is categorized as inadequate DLS between 0-<30 points, limited DLS between 30-<36 points, adequate DLS between 36-<42 points, and excellent DLS between 42-50 points. As the scores increase in the scale, the disaster literacy level of the participant increases.
Nurses' Perception of Disaster Preparedness Scale | 14 weeks
  This scale, which contains 20 items in total, consists of three sub-dimensions.The five-point Likert type scale includes the options "1-Strongly disagree, 2-Disagree, 3-Somewhat agree, 4-Agree, 5-Strongly agree" for rating. The higher the score obtained from the scale, the higher the perception of disaster preparedness.

CONTACTS AND LOCATIONS:
Overall Officials: özüm erkin, Ph.D, Principal Investigator — İzmir Democracy University
Locations (1):
- İzmir Democracy University, Izmir, Ege Bölgesi, Turkey (Türkiye)